CLINICAL TRIAL: NCT05345821
Title: Post-market Monitoring and Control of Safety and Efficacy of Silimed® Breast Implants with Smooth Surface (STEPS S)
Brief Title: An Analysis of Adverse Events and Satisfaction Outcomes of Women Who Underwent Primary and Secondary Breast Augmentation Using Silimed® Breast Implants with Smooth Surface
Acronym: STEPS S
Status: Recruiting | Type: Observational
Sponsor: Silimed Industria de Implantes Ltda (Industry)
Collaborators: Centro Universitário Saúde ABC (Other)
Responsible Party: Sponsor
Other Study IDs: 6001022
Record Dates: First submitted 2022-04-20; First posted 2022-04-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Breast Implant; Complications; Quality of Life; Satisfaction; Safety and Performance
Keywords: Breast Implant; satisfaction; qualify of life; smooth surface; post-market; safety; efficacy
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- primary augmentation group: Women undergoing primary breast augmentation with Silimed® smooth surface Breast Implant.
- secondary (revision) augmentation group: Women undergoing secundary or revision breast augmentation with Silimed® smooth surface Breast Implant.

SUMMARY:
The study investigates the safety and performance of Silimed® brand smooth surface breast implants in women born with indication for primary and secondary (revision) augmentation to be followed up for 10 years. The safety of the smooth-surfaced Silimed® implant will be evaluated by estimating known and unexpected short-term and long-term risk/adverse event rates through patient reports of adverse events after implantation. The performance of using Silimed® brand smooth surface breast implants will be evaluated by evaluating satisfaction and quality of life after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Female at birth
* Be 18 years of age or older
* Have a complaint of hypomastia
* Have an indication for breast augmentation with silicone implants
* Ability to comply with the protocol throughout the follow-up period.

Exclusion Criteria:

* Replacement of breast implants due to a complication
* Breast reconstruction in at least one breast
* Informed pregnancy or breastfeeding at the time of inclusion
* Sequelae of mastopexy
* Ptosis requiring mastopexy
* Breast changes or lumps rated BI-RADS 3 or higher on preoperative ultrasound or mammograms
* Advanced fibrocystic disease at the time of implantation
* Neoplasia of any type not yet treated or undergoing treatment at the time of implantation, - Active infection not yet treated or undergoing treatment at any site at the time of implantation
* Report or record of adverse reactions or intolerance to silicone prior to implantation
* Report or record of immune diseases affecting the active or undergoing treatment (e.g. lupus erythematosus, discoid lupus, scleroderma, etc.) at the time of implantation
* Signs of inflammation of the breast or implant site at the time of implantation
* Increased risk of post-implantation complications -immediate surgical complications caused by illicit drug use or medication use
* Having participated in another clinical trial within 6 months prior to implant placement
* Any other condition which, based on the opinion of the investigator or designee, may prevent the provision of informed consent, make study participation unsafe, compromise protocol adherence, complicate the interpretation of study outcome data, or otherwise interfere with the achievement of study objectives

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Born females with indication of primary and secondary augmentation (revision).
Sampling Method: Probability Sample
Enrollment: 384 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Expected Adverse Events | Every three years over the 10-year duration of the study
  Estimate the known short-term and long-term risk / adverse event rate for breast implant with smooth surface Silimed®
Unexpected Adverse Events | Every three years over the 10-year duration of the study
  Estimate the unknown short-term and long-term risk / adverse event rate for breast implant with smooth surface Silimed®

SECONDARY OUTCOMES:
Patient's Satisfaction in Relation to Aesthetic Result | Every three years over the 10-year duration of the study
  Estimate the performance of Silimed® breast implant with smooth surface through the satisfaction of the patient regarding the aesthetic result after breast augmentation. The assessment of patient's satisfaction will be done by means of a likert scale, where the following satisfaction options can be selected: 1 = definitely satisfied, 2 = satisfied, 3 = slightly satisfied, 4 = slightly dissatisfied and 5 = definitely unsatisfied.
Patient's Satisfaction in General | Every three years over the 10-year duration of the study
  Estimate the performance of Silimed® breast implants with smooth surface after breast augmentation by means of a questionnaire, the Breast Self-Assessment Questionnaire (BEQ-Brazil), which consist of 55 questions related to satisfaction and comfort with the overall appearance of the breasts.
Evaluator's Satisfaction in Relation to Aesthetic Result | Every three years over the 10-year duration of the study
  Estimate the performance of Silimed® breast implant with smooth surface througt the satisfaction of the evaluator regarding the aesthetic result after patient's breast augmentation. The assessment of evaluator's satisfaction will be done by means of a likert scale, where the following satisfaction options can be selected: 1 = definitely satisfied, 2 /= satisfied, 3= slightly satisfied, 4 = slightly dissatisfied and 5 = definitely unsatisfied.
Patient's Quality of Life | Every three years over the 10-year duration of the study
  Estimate the performance of Silimed® breast implant with smooth surface through the quality of life of the patient after breast augmentation. The assessment of patient's quality of life will be done by means of the Rosemberg Global Self-Esteem Scale, in order to evaluate the overall self-esteem of the sample.

CONTACTS AND LOCATIONS:
Overall Officials: André Luiz P de Freitas, Principal Investigator — Fundação do ABC - Centro Universitário FMABC
Locations (1):
- Fundação do ABC - Centro universitário FMABC, Santo André, São Paulo, Brazil